CLINICAL TRIAL: NCT06325189
Title: Effects of Aerobic Interval Training on Fatigue Level and Functional Performance in Post Angioplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec-42336
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease
Keywords: Angioplasty; Coronary Artery Disease; Fatigue; Recovery of Function; Rehabilitation
MeSH Terms: conditions — Coronary Artery Disease; Fatigue

STUDY DESIGN:
Intervention Model Description: In this parallel-group randomized controlled trial (RCT), post-angioplasty patients will be assigned to either the control group (receiving standard medication) or the experimental group (receiving medication along with aerobic interval training). The study aims to evaluate the impact of aerobic interval training on fatigue levels and functional performance in these patients.
Who Masked: Outcomes Assessor
Masking Description: The study was single-blinded, as assessors of the study were kept blind to the intervention group to which the participant was allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication alone (No Intervention): Participants in this arm will not receive any specific intervention. They will only receive standard care medications after angioplasty. No additional treatments or therapies will be administered.
- Aerobic Interval Training and medication (Experimental): In this arm, participants will receive the intervention. The intervention consists of aerobic interval training in addition to medication.
  Interventions: Other: Aerobic Interval Training

INTERVENTIONS:
Other: Aerobic Interval Training — Aerobic interval training is a cardiovascular exercise that involves short bursts of high-intensity activity followed by a brief rest or low-intensity exercise. It improves cardiovascular fitness, increases lung capacity, and enhances cardiovascular endurance. It also leads to higher calorie expenditure and time efficiency, allowing for faster fitness goals.
  Arms: Aerobic Interval Training and medication

SUMMARY:
The goal of this randomized controlled trial is to determine the effects of aerobic interval training on levels of tiredness and functional performance in post-angioplasty patients. The main question it aims to answer is:

Does aerobic interval training reduce fatigue and improve functional performance compared to medication alone in post-angioplasty patients?

Participants will:

Be randomly assigned to either the control group (medication) or the experimental group (medication + aerobic interval training) Perform aerobic interval training for 30 minutes, three times a week, for six weeks (experimental group only) Complete pre and post-intervention assessments using the fatigue severity scale, the 6-minute walk test, and the one minute sit to stand test Researchers will compare the two groups to see if aerobic interval training leads to significant improvements in fatigue levels and functional performance.

DETAILED DESCRIPTION:
The study is a randomized controlled trial that aims to evaluate the effects of aerobic interval training (AIT) on fatigue level and functional performance in post-angioplasty patients.

The study involves 47 participants who have undergone percutaneous coronary intervention (PCI) for coronary artery disease (CAD) and have completed phase 1 of cardiac rehabilitation.

The participants are divided into two groups: Group A receives medication only, and Group B receives medication plus AIT. The AIT consists of four sessions per week for four weeks, with each session lasting 40 minutes and alternating between high and low-intensity intervals.

The study hypothesizes that AIT will have a positive effect on fatigue level and functional performance in post-angioplasty patients, compared to medication alone.

The study uses descriptive statistics, paired t-tests, and independent t-tests to analyze the data and test the hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Patient with post angioplasty (having 1 or 2 stents)
* Patient who completed phase 1 cardiac rehabilitation
* Post coronary angioplasty patients 2 weeks of hospital discharge.

Exclusion Criteria:

* Patients with neurological disorders
* Patients with valvular and obstructive airway diseases.
* Patients with acute infections, malignancy
* Angioplasty complications such as arrhythmias, blood clots in-stent, and atrial fibrillations
* Patients with uncontrolled hypertension.
* Patients with uncontrolled diabetes.
* Presence of fracture.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | Baseline and four weeks
  This is a self-report measure that consists of nine items related to the level of fatigue and how it affects different tasks. The measure uses a seven-point scale, where 1 means strongly disagree and 7 means strongly agree. The lowest score that can be obtained is nine and the highest is 63. A higher score indicates a higher degree of fatigue and a greater impact on the person's activity. The measure is simple to comprehend and takes about eight minutes to complete.
Six Minute Walk Test | Baseline and four weeks
  Six Minute Walk Test is a measure of functional ability that is valid and reliable for the Phase II/III CR population. The 6-minute walk involves three walks, and a learning effect of six percent was observed. It is not known if this effect will persist in the long term. This test can be very useful for smaller CR centers that want to track functional progress but do not have the resources for conventional treadmill testing.
1 minute sit to stand: | Baseline and four weeks
  The 1-minute sit to stand test is a simple and quick fitness test that requires minimal equipment and space. It involves repeatedly standing up and sitting down on a chair for one minute and counting the number of repetitions. The test is reliable in measuring the functional capacity of cardiac patients, as it reflects their aerobic endurance and lower limb strength. The test can also help monitor the progress and response to cardiac rehabilitation programs.

CONTACTS AND LOCATIONS:
Overall Officials: Sumera Hamid, MS, Principal Investigator — Riphah International University
Locations (1):
- Gulab Devi Chest Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No